CLINICAL TRIAL: NCT05649202
Title: Hepatitis C in Prison: Study of Rapid Diagnosis and Treatment
Brief Title: Hepatitis C in Prison: Study of Screening and Rapid Treatment (HEPAPRIS)
Acronym: HEPAPRIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190948; 2019-A01418-49 (Other: ID-RCB Number)
Record Dates: First submitted 2022-10-10; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Chronic HIV Infection
Keywords: Hepatitis C; DAA; HCV Viral test; liver fibrosis
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All inmates entering the CPPLS: Patients with positive HCV serology
  Interventions: Other: Xpert® HCV Viral test; Other: FibroScan® test

INTERVENTIONS:
Other: Xpert® HCV Viral test — an additional sample of 5 ml of blood will be taken for real-time HCV PCR by Xpert®, in addition to the blood samples taken as part of routine care.
Other: FibroScan® test — A non invasive test made on a small area of skin coated with a gel
  Other Names: Presence of liver fibrosis Presence and importance of fat overload in the liver

SUMMARY:
Due to the high prevalence of HCV in prison and the risk of transmission between inmates, the management of hepatitis C and its treatment must be optimal following the recommendations of AFEF.

The purpose of this study is to assess the treatment starting delay from the date of incarceration of inmates with chronic HCV infection (hepatitis C).

DETAILED DESCRIPTION:
Detainees have specific health needs due to the high prevalence of several pathologies (HIV, HCV, tuberculosis, chronic diseases, addictions, psychiatric disorders associated in some cases with suicide attempts, etc.) and a degraded state of health. Detainees are frequently from the most disadvantaged social groups with low use of the health system prior to incarceration (drug users, people in precarious situations, migrants).

Although there is no data available in France about the incidence of HCV on inmates, several studies in France have documented exposure to the risk of transmission of hepatitis C through drug injection practices and sharing of injection equipment. The ANRS-Coquelicot survey focused at the national level on drug users attending the center of reception and support to risk reduction for drug users and the center of Care, Support and Prevention of addiction. In this survey, 12% of drug users reported injecting drugs during one of their incarcerations (61% of these users reported having been incarcerated at least once in their lifetime) and 30% reported sharing their injection equipment on that occasion [5]. These data have been confirmed in local studies that show practices in the reuse and share of injection equipment [6]. The PREVACAR survey showed that 18% of prison staff reported finding syringes in detention in the past 12 months [7]. These data are confirmed by the PRIDE survey in which one-third of caregivers reported having treated abscesses in inmates, probably related to injection practices [8].

Because of this high prevalence and the risk of transmission between inmates, treatment of hepatitis C in prison is highly recommended ([9], [10]).

However, there are difficulties in providing treatment. The main obstacle initially identified in 2014-15 was financial. Health care staff still face other challenges, particularly the difficulty of obtaining escorts in sufficient numbers to access technical trays and various consultations of local hospitals, with which the health units operate, and only 50% of medical extractions are carried out [12].

In addition, the conditions of medical extractions, with the almost systematic use of handcuffs and the frequent presence of supervisors at the consultation, while the assessment of the level of security to be implemented must be individualized (conditions noted by the evaluation report of the action plan and by the Controller of places of deprivation of liberty ( notice of 16/07/2015) often result in refusals on the part of detainees.

Another obstacle to the treatment of inmates is the short length of incarceration in a detention facility with an unknown release date for persons on a warrant of deposit. The most common causes of discontinued treatment is release (8%) (1.4%)) [13]. The rapid start of treatment for 8 or 12 weeks will prevent the interruption of most treatments. In addition, extra-carceral consultations are offered to all inmates leaving the CPPLS. This possibility is recorded in the welcome booklet and will be recalled when the treatment is started. These consultations are made by UCSA's general practitioners every morning from Tuesday to Friday from 8:30 a.m. to 12:30 p.m., without an appointment, at the Achard Pavilion Polyclinic at Cochin Hospital.

In accordance with the recommendations of the French Association for the Liver Study (AFEF) [14] this study proposes to optimize the medical care of prisoners with chronic HCV infection by reducing the time between diagnosis and on the way to AAD treatment, by using of the Xpert test® to determine the presence of viral RNA and also by extractions through a Fibroscan® to assess the degree of liver fibrosis.

This study proposes to determine the DAA (Direct-Acting Antiviral) treatment time frame defined by the time between the day of incarceration and the day of the start of DAA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>/= 18 years old),
* Persons detained at the Paris-La Santé Penitentiary Center (CPPLS) coming from the state of freedom or transferred from another penitentiary establishment
* Serology HCV positive

Exclusion Criteria:

* Major psychiatric disorders with loss of discernment
* Persons under guardianship or curatorship
* Persons not affiliated to a social security scheme

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons detained at the Paris-La Santé Penitentiary Center (CPPLS) from the state of liberty or transferred from another prison who have a positive HCV serology
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Delay to treat inmates with chronic HCV infection. | up to 8 days from incarceration
  The time frame for Direct-Acting Antiviral (DAA) treatment is defined by the time between the day of incarceration and the day of the DAA started.

SECONDARY OUTCOMES:
Describe the epidemiological data of the prison population of the Paris-La Santé Penitentiary Center (CPPLS) with positive HCV serology | At the inclusion
  Proportion of patients with positive HCV serology and description of clinical characteristics : age, transmission mode, co-infections (HIV, HBV) and comorbidities (alcohol, obesity, diabetes, renal failure), history of anti-HCV treatment.
Evaluate the rate of positive viral loads and describe the HCV genotypes in positive patients | At the inclusion
  Proportion of patients with a positive viral load by Xpert® HCV Viral test and proportion of the different HCV genotypes represented
Evaluate liver fibrosis of inmates with a positive HCV viral load | At the inclusion
  Proportion of patients with liver fibrosis assessed by FibroScan® test (level F1, F2, F3, F4) among patients with positive HCV viral load
Evaluate the cure rate at 12 weeks after the end of treatment | 12 weeks after the end of treatment
  * Proportion of patients with a negative HCV viral load at 12 weeks after stopping treatment
  * Cures defined as an undetectable viral load 12 weeks after stopping treatment
  * Duration of hepatitis C treatment

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ANDREW SILBERMANN, MsD, Principal Investigator — APHP
Locations (1):
- Internal Medicine Service, Cochin Hospital (Consultation and Ambulatory Care Unit (UCSA) within the Paris-La Santé Penitentiary Center (CPPLS)), Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiron E, Jauffret-Roustide M, Le Strat Y, Chemlal K, Valentin MA, Serre P, et al. Prévalence de l'infection par le VIH et le virus de l'hépatite C chez les personnes détenues en France. Résultats de l'enquête Prévacar 2010. Bull Epidemiol Hebd 2013 ; 35-36 : 445-50.
- [Background] Semaille C, Le Strat Y, Chiron E, Chemlal K, Valantin MA, Serre P, Cate L, Barbier C, Jauffret-Roustide M; Prevacar Group. Prevalence of human immunodeficiency virus and hepatitis C virus among French prison inmates in 2010: a challenge for public health policy. Euro Surveill. 2013 Jul 11;18(28):20524. doi: 10.2807/1560-7917.es2013.18.28.20524. PMID 23870097
- [Background] Jauffret-Roustide M, Le Strat Y, Couturier E, Thierry D, Rondy M, Quaglia M, Razafandratsima N, Emmanuelli J, Guibert G, Barin F, Desenclos JC. A national cross-sectional study among drug-users in France: epidemiology of HCV and highlight on practical and statistical aspects of the design. BMC Infect Dis. 2009 Jul 16;9:113. doi: 10.1186/1471-2334-9-113. PMID 19607712
- [Background] Sannier O, Verfaillie F, Lavielle D. [Risk reduction and drug use in detention: study about the detainees of Liancourt Penitentiary]. Presse Med. 2012 Jul;41(7-8):e375-85. doi: 10.1016/j.lpm.2011.12.015. Epub 2012 Mar 2. French. PMID 22386285
- [Background] Chemlal K, Bouscaillou J, Jauffret-Roustide M, Semaille C, Barbier C, Michon C, et al. Offre de soins en milieu carcéral en France : infection par le VIH et les hépatites. Enquête Prévacar, 2010. Bull Epidemiol Hebd 2012 ; 10-11 : 131-34.
- [Background] Michel L, Lions C, Van Malderen S, Schiltz J, Vanderplasschen W, Holm K, Kolind T, Nava F, Weltzien N, Moser A, Jauffret-Roustide M, Maguet O, Carrieri PM, Brentari C, Stover H. Insufficient access to harm reduction measures in prisons in 5 countries (PRIDE Europe): a shared European public health concern. BMC Public Health. 2015 Oct 27;15:1093. doi: 10.1186/s12889-015-2421-y. PMID 26507505
- [Background] Circulaire DGOS/R1/R4/DSS/1A/1C/2A n° 2015-148 du 29 avril 2015 relative à la facturation des AAD pour les patients pris en charge en ambulatoire dans des unités sanitaires en milieu pénitentiaire. http://social-sante.gouv.fr/fichiers/bo/2015/15-06/ste_20150006_0000_0065.pdf
- [Background] Brahmy B. [Difficulties medical care of persons placed under hand of justice]. Rev Prat. 2013 Jan;63(1):93-6. French. PMID 23457838
- [Background] Juan Jd, de la Hoya PS, Marco A, Anton JJ, Faraco I, Yllobre C, Pozo E, Hoyos C. Multicenter study on the discontinuation and efficacy of chronic hepatitis C treatment in the Spanish penitentiary population (EPIBAND study). Eur J Gastroenterol Hepatol. 2014 Oct;26(10):1083-9. doi: 10.1097/MEG.0000000000000163. PMID 25076064
- [Background] Lamoury FMJ, Bajis S, Hajarizadeh B, Marshall AD, Martinello M, Ivanova E, Catlett B, Mowat Y, Marks P, Amin J, Smith J, Ezard N, Cock V, Hayllar J, Persing DH, Kleman M, Cunningham P, Dore GJ, Applegate TL, Grebely J; LiveRLife Study Group. Evaluation of the Xpert HCV Viral Load Finger-Stick Point-of-Care Assay. J Infect Dis. 2018 May 25;217(12):1889-1896. doi: 10.1093/infdis/jiy114. PMID 29534185
- [Background] McHugh MP, Wu AHB, Chevaliez S, Pawlotsky JM, Hallin M, Templeton KE. Multicenter Evaluation of the Cepheid Xpert Hepatitis C Virus Viral Load Assay. J Clin Microbiol. 2017 May;55(5):1550-1556. doi: 10.1128/JCM.02460-16. Epub 2017 Mar 8. PMID 28275079
- [Background] Afdhal NH, Bacon BR, Patel K, Lawitz EJ, Gordon SC, Nelson DR, Challies TL, Nasser I, Garg J, Wei LJ, McHutchison JG. Accuracy of fibroscan, compared with histology, in analysis of liver fibrosis in patients with hepatitis B or C: a United States multicenter study. Clin Gastroenterol Hepatol. 2015 Apr;13(4):772-9.e1-3. doi: 10.1016/j.cgh.2014.12.014. Epub 2014 Dec 18. PMID 25528010
- See also: Related Info — http://www.justice.gouv.fr/prison-et-reinsertion-10036/la-vie-en-detention-10039/une-journee-type-en-prison-12005.html
- See also: Related Info — https://solidarites-sante.gouv.fr/IMG/pdf/rapport_.pdf